CLINICAL TRIAL: NCT00409032
Title: A Dose-response Study With Strontium Malonate in Postmenopausal Women. A 12 Week, Multi National, Double Blind, Randomized, 5 Arms, Parallel Group Placebo Controlled Open Label Active Controlled, Phase II Study With 3 Dose Levels of Strontium Malonate and Protelos Within Post Menopausal Women With a BMDT-score Below -1
Brief Title: A Dose-response Study With Strontium Malonate in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osteologix (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NBS-C03-OP
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Osteoporosis
Keywords: osteoporosis; BMD; CTX; Post menopausal; strontium; bone turnover; clinical development
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: Strontium malonate

SUMMARY:
The primary objective of the study is to compare dose-response effect of three dose levels of strontium malonate to placebo on bone resorption quantified by S-CTX-1 following 12 weeks of treatment.

DETAILED DESCRIPTION:
275 post menopausal women are treated with either 750 mg strontium malonate, 1000 mg strontium malonate, 2000 mg strontium malonate, 2 g Protelos® or placebo.

Patients are treated for 12 weeks. A follow up period of 4 weeks is planned for the main study and a follow up period of 8 weeks is planned for approximately 20% of the patients to follow post treatment CTX-1 activity.

Apart from S-CTS-1 also response on other bio markers are evaluated as well as BMD.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (at least 12 months since last menstruation).
* BMD (L2-4) T-score between -1 and -3 (at least 20% of the enrolled patients must have a BMD (L2-4) T-score below -2,5).
* 50 years of age.
* BMI<30 kg/m2.
* Total S-Ca level within normal range.
* Ability to read and understand the information given.
* The patient has signed an informed consent form according to ICH E6 and local requirements before any study specific procedure is carried out.
* Ability to comply with study procedures.

Exclusion Criteria:

* History of prior fragility fracture (any fracture in wrist, hip or spine appearing after 40 years of age).
* History of alcohol or drug abuse.
* Metabolic bone disease (e.g. pagets disease, bone cancer).
* History of VTE/DVT.
* History of kidney transplant.
* Bilateral oophorectomy.
* Relevant and treated reduced kidney or liver function.
* Any malignancy within the last 5 years (except basal cell carcinoma)
* Any chronic condition likely to affect absorption (e.g. Crohns disease, gluten enteropathy).
* Known genetic pre-disposition to VTE/DVT
* Known hypersensitivity to any of the active substances or excipients.
* 25-OH-vitamin D level below 25 nmol/L
* Any previous treatment with bisphosphonates, Strontium or fluoride.
* Treatment during the last 3 months affecting calcium balance or bone metabolism (e.g. thiazides, corticosteroids, calcitonin, HRT, SERMs, PTH, phosphorus).
* Treatment during the last week with tetracycline, ciprofloxacin or loop diuretics.
* PTH out of normal range
* Use of any drug known to influence the coagulation process (aspirin and other NSAID allowed)
* Prothrombin time out of normal range (sec or INR)
* Inclusion in another clinical study within 30 days before randomization or during this study

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
CTX-1

SECONDARY OUTCOMES:
Other bio markers, BMD

CONTACTS AND LOCATIONS:
Overall Officials: Richard Eastell, Professor, M.D., Principal Investigator — University of Sheffield, Metabolic Bone Centre, Northern General Hospital, Sheffield S5 7AU, United Kingdom
Locations (9):
- Denmark (2):
  - PhaseOneTrials, Hvidovre
  - Odense University Hospital, Odense
- United Kingdom (7):
  - Medinova Clinic, Northwood, Middlesex
  - Synexus Wales Clinical Research Centre, Cardiff
  - Synexus Scotland Clinical Research Centre, Glasgow
  - Synexus Limited Reading Clinical Research Centre, Reading
  - University of Sheffield, Sheffield
  - Synexus Crosby Clinical Research Centre, Waterloo
  - Synexus Wigan Clinical Research Centre, Wigan

REFERENCES:
- See also: Related Info — http://www.osteologix.com